CLINICAL TRIAL: NCT00036712
Title: A Multiinstitutional Trial To Evaluate The Prophylactic Use Of NASA-Developed Light Emitting Diodes For The Prevention Of Oral Mucositis In Bone Marrow Transplant Patients
Brief Title: Light-Emitting Diode Therapy in Preventing Mucositis in Children Receiving Chemotherapy With or Without Radiation Therapy Before Bone Marrow Transplantation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Harry T. Whelan, Medical College of Wisconsin Cancer Center
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Supportive Care
Other Study IDs: CDR0000069293; MCW-HRRC-28600; MCW-CHW-0070; NCI-V02-1699
Record Dates: First submitted 2002-05-13; First posted 2003-01-27 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2009-06

CONDITIONS: Chronic Myeloproliferative Disorders; Kidney Cancer; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms; Neuroblastoma; Oral Complications; Ovarian Cancer; Pain; Sarcoma
Keywords: recurrent childhood acute lymphoblastic leukemia; refractory multiple myeloma; recurrent childhood rhabdomyosarcoma; disseminated neuroblastoma; recurrent neuroblastoma; recurrent Wilms tumor and other childhood kidney tumors; recurrent childhood lymphoblastic lymphoma; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; recurrent childhood acute myeloid leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; primary myelofibrosis; childhood acute promyelocytic leukemia (M3); refractory hairy cell leukemia; oral complications; recurrent/refractory childhood Hodgkin lymphoma; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; pain; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; previously treated childhood rhabdomyosarcoma; childhood malignant ovarian germ cell tumor; childhood chronic myelogenous leukemia; atypical chronic myeloid leukemia, BCR-ABL1 negative; myelodysplastic/myeloproliferative neoplasm, unclassifiable; childhood myelodysplastic syndromes
MeSH Terms: conditions — Myeloproliferative Disorders; Kidney Neoplasms; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Neuroblastoma; Ovarian Neoplasms; Pain; Sarcoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Wilms Tumor; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Primary Myelofibrosis; Leukemia, Hairy Cell; Recurrence; Burkitt Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Ovarian Germ Cell Cancer; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative | interventions — Analgesia

INTERVENTIONS:
Procedure: management of therapy complications
Procedure: pain therapy

SUMMARY:
RATIONALE: Light-emitting diode (LED) therapy may be able to prevent mucositis of the mouth.

PURPOSE: Randomized phase II trial to determine the effectiveness of LED therapy in preventing mucositis of the mouth in children who are receiving chemotherapy with or without radiation therapy before donor bone marrow transplantation.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the incidence and severity of oral mucositis in children undergoing NASA-developed light-emitting diode (LED) therapy during a pre-transplantation myeloablative conditioning regimen (chemotherapy with or without radiotherapy) and continuing through the post-bone marrow transplantation (BMT) phase versus LED therapy during the post-BMT phase only.

OUTLINE: This is a randomized, double-blind, multicenter study. Patients are stratified according to participating center and cheek being treated (right vs left). Patients are randomized to 1 of 2 schedules of light-emitting diode (LED) therapy.

* Arm I: Patients undergo LED therapy for 71 seconds once daily beginning on day 1 of the myeloablative conditioning regimen comprising chemotherapy with or without radiotherapy and continuing for 14 days after bone marrow transplantation (BMT).
* Arm II: Patients undergo LED therapy as in arm I beginning on the day of BMT (day 0) and continuing for 14 days after BMT.

Photographs are taken of the right and left buccal mucosa at baseline and then every 3 days beginning on day 1 of LED therapy.

Pain and xerostomia are assessed using the Wong-Baker "smiley-face" pain scale at baseline and then periodically for 14 days after BMT.

Patients are followed monthly for 2 years.

PROJECTED ACCRUAL: A total of 80 patients (40 per arm) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients undergoing a myeloablative conditioning regimen comprising chemotherapy with or without radiotherapy prior to a first allogeneic bone marrow transplantation

PATIENT CHARACTERISTICS:

Age:

* 2 to 18

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Pulmonary:

* No pulmonary dysfunction that would increase significantly the risk of requiring intubation during the first 21 days after transplantation

Other:

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* No photophobia
* Must have emotional, cognitive, and mental maturity sufficient to tolerate light-emitting diode therapy application and oral examination without combativeness

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics

Surgery:

* Not specified

Other:

* No concurrent medication that may cause epidermal or ocular photosensitivity

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2002-01; Primary Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
Mean change in oral mucositis index (OMI) score from baseline to maximum score within 14 days posttransplant
Mean change in pain score from baseline to maximum score within 14 days posttransplant
Proportion of patients not experiencing ulcerative mucositis within the first 14 days posttransplant

SECONDARY OUTCOMES:
Time to heal

CONTACTS AND LOCATIONS:
Overall Officials: Harry T. Whelan, MD, Study Chair — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin, United States